CLINICAL TRIAL: NCT04019106
Title: Pharmacokinetics and Pharmacodynamics of Budesonide With Intratracheal Surfactant (BITS) Administration in Preterm Infants < 29 Weeks Gestational Age
Brief Title: Budesonide With Intratracheal Surfactants in Extremely Preterm Infants
Acronym: BITS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre, Winnipeg, Manitoba (Other); St. Boniface Hospital (Other); Manitoba Institute of Child Health (Industry); University of Utah (Other); Winnipeg Rh Institute Foundation Inc. (Unknown); BLES Biochemicals Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BITS-03
Record Dates: First submitted 2018-08-15; First posted 2019-07-15 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2018-08

CONDITIONS: Bronchopulmonary Dysplasia; Respiratory Distress Syndrome in Premature Infant
Keywords: Surfactant; Budesonide; Steroid; Intratracheal; Preterm; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome; Bovine Lipid Extract Surfactant
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Respiratory Distress Syndrome | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dosing Level 1 (Experimental): 0.0625 mg/kg Budesonide in bovine lipid extract surfactant (BLES)
  Interventions: Drug: Budesonide in bovine lipid extract surfactant (BLES)
- Dosing Level 2 (Experimental): 0.125 mg/kg Budesonide in bovine lipid extract surfactant (BLES)
  Interventions: Drug: Budesonide in bovine lipid extract surfactant (BLES)
- Dosing Level 3 (Experimental): 0.25 mg/kg Budesonide in bovine lipid extract surfactant (BLES)
  Interventions: Drug: Budesonide in bovine lipid extract surfactant (BLES)

INTERVENTIONS:
Drug: Budesonide in bovine lipid extract surfactant (BLES) — Budesonide in bovine lipid extract surfactant
  Other Names: Pulmicort respule; BLES

SUMMARY:
This is a phase I/II trial in preterm infants aimed at identifying the optimal dose of budesonide with bovine lipid extract surfactant as vehicle for intratracheal administration.

DETAILED DESCRIPTION:
Premature infants of gestational age less than 29 weeks with respiratory distress syndrome and clinical indication for surfactant administration will be recruited for this Phase I/II open-label study.

A total of 30 subjects will be recruited from 2 neonatal intensive care units:

1. Children's Hospital-Health Sciences Centre (HSC), Winnipeg
2. St. Boniface General Hospital, Winnipeg, MB

3 groups of 10 infants each will receive single dose of intratracheal budesonide (0.0625 mg/kg, 0.125 mg/kg, and 0.25 mg/kg) with BLES surfactant (5 ml/kg). PK/PD analysis will be done using clinical parameters, serum biomarkers, tracheal aspirate biomarkers and plasma budesonide levels obtained at fixed intervals.

The duration of subject participation will involve 12-17 weeks for the clinical intervention, depending on gestational age at birth and discharge date. Participants will be followed until 40 weeks or discharge, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infant born between 23 and 28+6 weeks of GA
2. Infant diagnosed with RDS according to clinical protocol criteria
3. Able to adhere to surfactant administration protocol
4. The patient is born in the study centre.
5. Subject's parent(s)/legal guardian(s) has provided signed and dated informed consent and authorization to use protected health information, as required by national and local regulations.
6. In the investigator's opinion, the subject's parent(s)/legal guardian(s) understand(s) and can comply with protocol requirements, instructions, and protocol-stated restrictions, and is likely to complete the study as planned.

Exclusion Criteria:

1. Older than five days at inclusion.
2. Presence of known clinically significant congenital heart disease or other major congenital malformation
3. Subjects with clinically significant laboratory abnormalities which are deemed by the investigator to represent a safety risk to participation in this study. Other laboratory parameters outside the reference range for the subject's age may be included if the investigator considers the abnormalities unlikely to introduce additional risk factors and will not interfere with data interpretation.

Ages: 1 Hour to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-10-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from serial budesonide levels | At 24 hour time point following dosing
  Blood samples will be drawn from patients to determine the serum budesonide levels to determine the area under the curve

SECONDARY OUTCOMES:
Bronchopulmonary Dysplasia free survival | at 36 weeks PMA or discharge, whichever comes first
  NICHD criteria will be used to diagnose and grade the infants for presence of BPD.
Neonatal Mortality | up to 40 weeks PMA or discharge, whichever comes first
  Survival of the infants
Concentration of Inflammatory Biomarkers in Tracheal Aspirates | Baseline, 24 hours, 48 hours,1 week, 4 weeks and 36 weeks Gestational Age
  Tracheal aspirates will be centrifuged to isolate a large aggregate surfactant fraction that will be assayed for both phospholipid (surfactant recovery) and total protein concentration. The supernatant fraction after surfactant isolation will be assayed for total protein, and selected cytokines (IL-1 β, IL-6, IL-8, IL-10, CCL2 and TNF-ɑ)
Concentration of Inflammatory Biomarkers in Serum | Baseline, 24 hours, 48 hours and 1 week.
  Cytokines IL-1 β, IL-6, IL-8, IL-10, CCL2 and TNF-ɑ will be analyzed in serum samples obtained from the infants following BITS administration using commercially available ELISA kits.
Duration of Hospital Stay | from day 0 (birth date) to 40 weeks
VentilationStrategy | till 36 weeks PMA or discharge, whichever comes first
  Duration and modality of ventilation used in the preterm infants
Respiratory Severity Score | at baseline and till 36 weeks PMA or discharge, whichever comes first
  The product of Fraction of inspired oxygen and mean airway pressure will be used to estimate the respiratory severity score
Duration of Supplemental Oxygen | till 36 weeks PMA or discharge, whichever comes first
Level of Supplemental Oxygen Administered | at baseline and at 36 week Post menstrual age or discharge, whichever comes first
  the concentration of supplemental oxygen given at discharge or 36 weeks PMA compared to baseline.
Presence of Respiratory Support | at 36 week Post menstrual age or discharge, whichever comes first
  the presence or absence of any method of respiratory support at discharge or 36 weeks PMA compared to baseline.
Percentage of Participants with Pulmonary Hemorrhage | at baseline and 48 hours after budesonide with surfactant administration
  Clinical signs of pallor, cyanosis, bradycardia, apnoea and blood gas changes. Radiographic evidences of patchy infiltrates to complete opacification of lung fields.
Percentage of Participants with Hypothalamic pituitary axis (HPA) suppression | at 0 and 24 hours after dosing
  Cortisol levels will be measured
Percentage of Participants with Pneumothorax on Chest X-ray | at baseline and 48 hours after budesonide with surfactant administration
  Identified in X-ray as hyperlucent shadow outside the lungs without pulmonary vascular markings, with or without mediastinal shift
Percentage of Participants with Spontaneous Intestinal Perforation (SIP) on abdominal X-ray | at baseline and 48 hours after budesonide with surfactant administration
  Abdominal X-ray showing presence of free air. Presence or absence of SIP will be compared across the 3 dosing groups and within the dosing groups.
Percentage of Participants with Intra-ventricular Hemorrhage | at baseline and 48 hours after budesonide with surfactant administration
  presence or absence of will be compared across the 3 dosing groups and within the dosing groups.
Percentage of Participants with Sepsis | at baseline and till 36 weeks PMA or discharge, whichever comes first
  As per the third international consensus definitions for sepsis and septic shock (Sepsis-3)
Percentage of Participants with Necrotising Enterocolitis (NEC) | 48 hours after budesonide with surfactant administration
  presence or absence of NEC will be compared across the 3 dosing groups and within the dosing groups.
Percentage of Participants with Severe Retinopathy at Prematurity | baseline and 48 hours after budesonide with surfactant administration
  retinopathy of ≥grade III will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Geert W 't Jong, MD, Ph.D, Principal Investigator — Children's Hospital Research Institute of Manitoba
Locations (2):
- Canada (2):
  - Children's Hospital-Health Science Centre, Winnipeg, Manitoba
  - St. Boniface General Hospital, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: Undecided